CLINICAL TRIAL: NCT07044102
Title: The Effect of Continuous Low Tidal Volume Ventilation During Cardiopulmonary Bypass on Renal Resistive Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Esra GÖGER, Specialist Doctor, MD Anesthesiology and Reanimation, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bypass surgery
Record Dates: First submitted 2025-06-23; First posted 2025-06-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: participants are randomized in a parallel design to receive either continuous low tidal volume ventilation or conventional ventilation during cardiopulmonary bypass
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Undergoing Low Tidal Volume Ventilation During CABG (Experimental): patients undergoing coronary artery bypass grafting receive continuous low tidal volume ventilation during cardiopulmonary bypass
  Interventions: Other: Patients Undergoing Low Tidal Volume Ventilation During CABG
- Patients Managed With Apneic Ventilation During Cardiopulmonary Bypass" (Active Comparator): patients undergoing coronary artery bypass grafting are managed with apnea ventilation during cardiopulmonary bypass
  Interventions: Other: Patients Undergoing Apneic Ventilation During CABG

INTERVENTIONS:
Other: Patients Undergoing Low Tidal Volume Ventilation During CABG — Postoperative Evaluation of Renal Resistive Index Using Doppler Ultrasound After Cardiopulmonary Bypass
  Arms: Patients Undergoing Low Tidal Volume Ventilation During CABG
Other: Patients Undergoing Apneic Ventilation During CABG — Postoperative Evaluation of Renal Resistive Index Using Doppler Ultrasound After Cardiopulmonary Bypass"
  Arms: Patients Managed With Apneic Ventilation During Cardiopulmonary Bypass"

SUMMARY:
Postoperative acute kidney injury following cardiopulmonary bypass surgery represents a significant barrier to patient recovery and is closely associated with increased postoperative morbidity and mortality. Studies have shown that the incidence of AKI aftercardiopulmonary bypass surgeryranges between 5% and 30%.

The Renal Resistive Index, measured by Doppler ultrasonography, is an increasingly utilized parameter that provides valuable insights into renal hemodynamics and vascular resistance. A normal RRI is typically below 0.70; elevated values may indicate increased renal vascular resistance or microvascular damage. Bossard et al. demonstrated that increased RRI in the early postoperative period is associated with the development of AKI. Early evaluation of renal blood flow thus facilitates prompt detection of AKI. Both preoperative and postoperative RRI measurements are considered useful tools for identifying early renal dysfunction. Monitoring RRI before and after CABG may provide critical information for preventing postoperative renal complications.

DETAILED DESCRIPTION:
Postoperative acute kidney injury following cardiopulmonary bypass surgery represents a significant barrier to patient recovery and is closely associated with increased postoperative morbidity and mortality. Studies have shown that the incidence of AKI after CABG ranges between 5% and 30%.

The Renal Resistive Index, measured by Doppler ultrasonography, is an increasingly utilized parameter that provides valuable insights into renal hemodynamics and vascular resistance. A normal RRI is typically below 0.70; elevated values may indicate increased renal vascular resistance or microvascular damage. Bossard et al. demonstrated that increased RRI in the early postoperative period is associated with the development of AKI. Early evaluation of renal blood flow thus facilitates prompt detection of AKI. Both preoperative and postoperative RRI measurements are considered useful tools for identifying early renal dysfunction. Monitoring RRI before and after CABG may provide critical information for preventing postoperative renal complications.In recent years, significant advancements have been made in both surgical and anesthetic techniques in cardiac surgery. During CABG, the commonly used ventilation strategy during cardiopulmonary bypass is apneic ventilation. However, low tidal volume ventilation has been proposed as an alternative, with a growing body of literature supporting its use. LTV has been associated with reduced postoperative pulmonary complications, earlier extubation, and prevention of atelectasis and pulmonary edema.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac bypass surgery
* Male and female patients over 18 years of age
* Patients with an American Society of Anesthesiologists (ASA) physical status classification of II, III, or IV

Exclusion Criteria:

* Chronic renal failure requiring dialysis
* Patients requiring emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Renal resistive ındex | Postoperative 45 minutes
  Measurement of Changes in Renal Resistive Index Associated With Low Tidal Volume and Apneic Ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)